CLINICAL TRIAL: NCT00686725
Title: A Clinical Study of Standard TEMODAL® Regimen Versus Standard Regimen Plus Early Post-Surgery TEMODAL® Chemotherapy in Treatment on Patients With Newly Diagnosed Glioblastoma Multiforme (GBM)
Brief Title: Standard Temodal (Temozolomide) Regimen Versus Standard Regimen Plus Early Postsurgery Temodal for Newly Diagnosed Glioblastoma Multiforme (Study P05572)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P05572
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Results first posted 2013-04-04 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Temozolomide + Radiation (Active Comparator): Standard therapy regimen:
  Treatment will start 4 weeks after surgery. Temozolomide will be administered concomitantly with radiotherapy, at 75 mg/m^2/day orally for 42 days. Four weeks after completing concomitant radiotherapy, temozolomide will be administered for an additional six cycles. Each cycle will last 28 days, and temozolomide will be administered once daily from Day 1 to Day 5 of each cycle. The dose of temozolomide in the first cycle will be 150 mg/m^2/day, and may be increased to 200 mg/m^2/day for Cycle 2 and subsequent cycles depending on nonhematological toxicity observed and neutrophil and platelet count values. Capsules containing 20 mg or 100 mg of temozolomide will be used.
  Radiotherapy will be administered in combination with temozolomide. Radiotherapy will be administered for a total daily dose of 60 Gy in 30 fractions, 5 days a week for 6 weeks.
  Interventions: Drug: Temozolomide; Radiation: Radiotherapy
- Temozolomide alone, then Temozolomide + Radiation (Experimental): Early postsurgery temozolomide chemotherapy plus standard regimen:
  Treatment with temozolomide alone will start 2 weeks after surgery at 75 mg/m^2/day orally for 14 days. Then, starting on Day 29 after surgery, temozolomide will be administered according to standard treatment as described for the temozolomide + radiation arm (standard therapy regimen).
  Radiotherapy will be administered in combination with temozolomide. Radiotherapy will be administered for a total daily dose of 60 Gy in 30 fractions, 5 days a week for 6 weeks.
  Interventions: Drug: Temozolomide; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Temozolomide
  Other Names: Temodal; Temodar; SCH 052365
Radiation: Radiotherapy
  Other Names: Irradiation; radiation therapy

SUMMARY:
The primary purpose of the study is to evaluate the efficacy and safety of early postsurgery temozolomide chemotherapy followed by the standard temozolomide regimen, compared to the standard regimen alone, for the treatment of patients with newly diagnosed glioblastoma multiforme.

ELIGIBILITY:
Inclusion Criteria:

Only the patients who meet all these criteria can be enrolled in the study:

* Patients with prior histological confirmation of newly diagnosed primary glioblastoma multiforme in supratentorial cerebral hemisphere.
* Gross total resection or partial resection (imaging) >70%.
* At least be capable to obtain a tissue sample for MGMT analysis during surgery.
* Chemo-radiotherapy to be expected from Week 5 (Day 29) after surgery.
* Age >=18 and <=70 years.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* Life expectancy >=9 months.
* Laboratory test values must satisfy the following criteria:

  * absolute neutrophil count >=1.5 x 10^9/L;
  * platelet count >=100 x 10^9/L;
  * hemoglobin >=80 g/L;
  * blood urea nitrogen and creatinine < 1.5 x upper limit of normal value (ULN);
  * total bilirubin and direct bilirubin < 1.5 x ULN;
  * alanine aminotransferase and aspartate aminotransferase < 3 x ULN;
  * alkaline phosphatase < 2 x ULN.
* Patients must be willing to provide written informed consent.
* Patients of child-bearing potential (including female subjects and the female partners of male subjects) must use an effective method of contraception.

Exclusion Criteria:

Patients will not be enrolled if any of the following criteria apply:

* Patient with previous or current malignancies (except melanoma) at other sites, unless disease free for at least 3 years.
* Patient who received chemotherapy, radiotherapy for study indication, or other medications for antitumor indication prior to surgery.
* Patient with recurrent or multiple malignant glioma (including gliomatosis cerebri).
* Patient with metastatic lesions at the subtentorial or outside of calvaria.
* Patient who received chemotherapy or radiotherapy sensitizers for head or neck tumor.
* Patient who received radiotherapy at head or neck which leads to radiotherapy domain overlapping.
* Patient with acute infections requiring intravenous antibiotics.
* Frequent vomiting or medical condition that could interfere with oral medication intake (eg, partial bowel obstruction).
* Known human immunodeficiency virus (HIV)-positive or acquired immune deficiency syndrome (AIDS)-related illness.
* Woman who is pregnant or breastfeeding.
* Patient with a history of hypersensitivity to temozolomide or other analogic alkylating agents.
* Patient with any other conditions under which investigators think the subject is not suitable for enrolment, such like having known that the subject may not have good compliance.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2008-06-24 (Actual); Primary Completion 2011-09-28 (Actual); Study Completion 2011-09-28 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Mao Y, Yao Y, Zhang LW, Lu YC, Chen ZP, Zhang JM, Qi ST, You C, Wang RZ, Yang SY, Zhang X, Wang JS, Chen JX, Yang QY, Shen H, Li ZY, Wang X, Ma WB, Yang XJ, Zhen HN, Zhou LF. Does Early Postsurgical Temozolomide Plus Concomitant Radiochemotherapy Regimen Have Any Benefit in Newly-diagnosed Glioblastoma Patients? A Multi-center, Randomized, Parallel, Open-label, Phase II Clinical Trial. Chin Med J (Engl). 2015 Oct 20;128(20):2751-8. doi: 10.4103/0366-6999.167313. PMID 26481741

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Temozolomide + Radiation | Temozolomide Alone, Then Temozolomide + Radiation
Started | 47 | 52
Completed | 1 (Completers were defined as those who completed the established treatment.) | 10 (Completers were defined as those who completed the established treatment.)
Not Completed | 46 | 42
Not completed — Adverse Event | 1 | 1
Not completed — Progressive Disease | 17 | 23
Not completed — Lost to Follow-up | 7 | 5
Not completed — Death | 6 | 3
Not completed — Withdrawal by Subject | 13 | 4
Not completed — Protocol Violation | 1 | 3
Not completed — Other | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Temozolomide + Radiation | Temozolomide Alone, Then Temozolomide + Radiation | Total
Number analyzed (Participants) | 47 | 52 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (10.12) | 48.5 (13.04) | 50.2 (11.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 20 | 33
  Male | 34 | 32 | 66
Region of Enrollment [Number; unit: participants]
  China | 47 | 52 | 99

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death.
  OS was calculated by the Kaplan-Meier method.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Temozolomide + Radiation | Temozolomide Alone, Then Temozolomide + Radiation
Number analyzed (Participants) | 47 | 52
months | 13.17 [11.14 to 18.76] | 17.58 [15.18 to 23.03]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the length of time from randomization to disease progression (the length of time during which the cancer did not get worse) or death.
  PFS was calculated by the Kaplan-Meier method.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Temozolomide + Radiation | Temozolomide Alone, Then Temozolomide + Radiation
Number analyzed (Participants) | 47 | 52
months | 10.38 [8.18 to 15.44] | 8.74 [6.41 to 14.85]

3. Secondary Outcome: Objective Tumor Assessment After Surgery: Overall Response
Description: Overall response was based on neuroimaging (magnetic resonance imaging [MRI]), clinical neurological examination, and steroid administration.
  It was assessed as follows:
  Complete Response (CR): Disappearance of all enhancing tumor (measurable
  or non-measurable), no corticosteroid use, and neurologically stable or
  improved.
  Partial Response (PR): ≥50% reduction in size of enhancing tumor
  (measurable or non-measurable) for any measurable lesions or definite
  improvement for any non-measurable lesions, corticosteroid dosage stable or
  reduced, and neurologically stable or improved.
  Progressive Disease (PD): ≥25% increase in contrast enhancement for any
  measurable lesions or definite worsening for any non-measurable lesions, or
  any new tumor on MRI scans, at an increased dose of corticosteroid, with or without neurologic progression. Clinical or radiological worsening resulting from other than tumor factors were excluded.
  Stable Disease (SD): All other situations.
Time Frame: Up to 2 years
Measure: Number; unit: participants
Arm/Group | Temozolomide + Radiation | Temozolomide Alone, Then Temozolomide + Radiation
Number analyzed (Participants) | 47 | 52
participants
  CR | 1 | 0
  PR | 0 | 0
  SD | 38 | 47
  PD | 3 | 4
  No overall response data available | 5 | 1

4. Secondary Outcome: Relationship Between O6-methylguanine-DNA Methyltransferase (MGMT) Status and Therapy Response: Overall Survival for the MGMT Positive Group
Description: MGMT was measured by immunohistochemistry (IHC).
  OS was defined as the length of time from the start of treatment that 1/2 of the participants were still alive.
  OS was calculated by the Kaplan-Meier method.
Time Frame: Up to 2 years
Population: Participants with enough tissue to perform MGMT analysis.
  Only MGMT-positive participants are included in this outcome measure. MGMT-negative participants are reported in outcome measure 5.
Measure: Median (Standard Deviation); unit: months
Arm/Group | Temozolomide + Radiation | Temozolomide Alone, Then Temozolomide + Radiation
Number analyzed (Participants) | 15 | 20
months | 14.4 (2.385) | 17.49 (1.491)
Statistical Analysis 1: Comparison: Temozolomide + Radiation vs Temozolomide Alone, Then Temozolomide + Radiation; Test type: Superiority or Other; p = 0.183, Log Rank

5. Secondary Outcome: Relationship Between MGMT Status and Therapy Response: Overall Survival for the MGMT Negative Group
Description: MGMT was measured by IHC.
  OS was defined as the length of time from the start of treatment that 1/2 of the participants were still alive.
  OS was calculated by the Kaplan-Meier method.
Time Frame: Up to 2 years
Population: Participants with enough tissue to perform MGMT analysis.
  Only MGMT-negative participants are included in this outcome measure. MGMT-positive participants are reported in outcome measure 4.
Measure: Median (Standard Deviation); unit: months
Arm/Group | Temozolomide + Radiation | Temozolomide Alone, Then Temozolomide + Radiation
Number analyzed (Participants) | 27 | 28
months | 13.81 (1.417) | 15.12 (1.171)
Statistical Analysis 1: Comparison: Temozolomide + Radiation vs Temozolomide Alone, Then Temozolomide + Radiation; Test type: Superiority or Other; p = 0.35, Log Rank

6. Secondary Outcome: Relationship Between MGMT Status and Therapy Response: Overall Survival Rate for the MGMT Positive Group
Description: MGMT was measured by IHC.
  OS rate was defined as the percentage of participants who were still alive 6, 12, & 18 months after starting study treatment.
  OS was calculated by the Kaplan-Meier method.
Time Frame: 6, 12, & 18 months
Population: Participants with enough tissue to perform MGMT analysis.
  Only MGMT-positive participants are included in this outcome measure. MGMT-negative participants are reported in outcome measure 7.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Temozolomide + Radiation | Temozolomide Alone, Then Temozolomide + Radiation
Number analyzed (Participants) | 15 | 20
percentage of participants
  6 months | 80.8 [42.3 to 94.9] | 89.2 [63.1 to 97.2]
  12 months | 69.3 [31.2 to 89.1] | 82.8 [55.4 to 94.2]
  18 months | 36.9 [6.5 to 69.6] | 66.2 [35.7 to 84.8]

7. Secondary Outcome: Relationship Between MGMT Status and Therapy Response: Overall Survival Rate for the MGMT Negative Group
Description: as for outcome 6
Time Frame: 6, 12, & 18 months
Population: Participants with enough tissue to perform MGMT analysis.
  Only MGMT-negative participants are included in this outcome measure. MGMT-positive participants are reported in outcome measure 6.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Temozolomide + Radiation | Temozolomide Alone, Then Temozolomide + Radiation
Number analyzed (Participants) | 27 | 28
percentage of participants
  6 months | 87.5 [66.1 to 95.8] | 95.8 [73.9 to 99.4]
  12 months | 57.7 [31.9 to 76.8] | 81.4 [57.5 to 92.6]
  18 months | 44.9 [21.1 to 66.3] | 26.7 [9.1 to 48.3]

8. Secondary Outcome: Relationship Between MGMT Status and Therapy Response: PFS for the MGMT Positive Group
Description: MGMT was measured by IHC.
  PFS: The length of time during and after treatment that a participant lived with the cancer but it does not get worse.
  PFS was calculated by the Kaplan-Meier method.
Time Frame: Up to 2 years
Population: Participants with enough tissue to perform MGMT analysis.
  Only MGMT-positive participants are included in this outcome measure. MGMT-negative participants are reported in outcome measure 9.
Measure: Median (Standard Deviation); unit: months
Arm/Group | Temozolomide + Radiation | Temozolomide Alone, Then Temozolomide + Radiation
Number analyzed (Participants) | 15 | 20
months | 10.04 (2.094) | 11.19 (1.882)
Statistical Analysis 1: Comparison: Temozolomide + Radiation vs Temozolomide Alone, Then Temozolomide + Radiation; Test type: Superiority or Other; p = 0.648, Log Rank

9. Secondary Outcome: Relationship Between MGMT Status and Therapy Response: PFS for the MGMT Negative Group
Description: as for outcome 8
Time Frame: Up to 2 years
Population: Participants with enough tissue to perform MGMT analysis.
  Only MGMT-negative participants are included in this outcome measure. MGMT-positive participants are reported in outcome measure 8.
Measure: Median (Standard Deviation); unit: months
Arm/Group | Temozolomide + Radiation | Temozolomide Alone, Then Temozolomide + Radiation
Number analyzed (Participants) | 27 | 28
months | 11.11 (1.441) | 10.46 (1.475)
Statistical Analysis 1: Comparison: Temozolomide + Radiation vs Temozolomide Alone, Then Temozolomide + Radiation; Test type: Superiority or Other; p = 0.915, Log Rank

ADVERSE EVENTS:
Description: Population is all treated participants.
Groups:
- Temozolomide Radiation: Standard therapy regimen: Treatment will start 4 weeks after surgery. Temozolomide will be administered concomitantly with radiotherapy, at 75 mg/m^2/day orally for 42 days. Four weeks after completing concomitant radiotherapy, temozolomide will be administered for an additional six cycles. Each cycle will last 28 days, and temozolomide will be administered once daily from Day 1 to Day 5 of each cycle. The dose of temozolomide in the first cycle will be 150 mg/m^2/day, and may be increased to 200 mg/m^2/day for Cycle 2 and subsequent cycles depending on nonhematological toxicity observed and neutrophil and platelet count values. Capsules containing 20 mg or 100 mg of temozolomide will be used. Radiotherapy will be administered in combination with temozolomide. Radiotherapy will be administered for a total daily dose of 60 Gy in 30 fractions, 5 days a week for 6 weeks.
- Temozolomide Alone, Then Temozolomide Radiation: Early postsurgery temozolomide chemotherapy plus standard regimen: Treatment with temozolomide alone will start 2 weeks after surgery at 75 mg/m^2/day orally for 14 days. Then, starting on Day 29 after surgery, temozolomide will be administered according to standard treatment as described for the temozolomide radiation arm (standard therapy regimen). Radiotherapy will be administered in combination with temozolomide. Radiotherapy will be administered for a total daily dose of 60 Gy in 30 fractions, 5 days a week for 6 weeks.
Arm/Group | Temozolomide Radiation | Temozolomide Alone, Then Temozolomide Radiation
Serious Adverse Events (participants affected / at risk) | 11/42 | 11/52
Other Adverse Events (participants affected / at risk) | 24/42 | 22/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temozolomide Radiation (N=42) | Temozolomide Alone, Then Temozolomide Radiation (N=52)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0)
DISEASE PROGRESSION (General disorders) | 3 (3) | 2 (2)
DISEASE RECURRENCE (General disorders) | 1 (1) | 0 (0)
HEPATIC FAILURE (Hepatobiliary disorders) | 1 (1) | 0 (0)
CENTRAL NERVOUS SYSTEM INFECTION (Infections and infestations) | 0 (0) | 1 (1)
LUNG INFECTION (Infections and infestations) | 0 (0) | 1 (1)
BRAIN HERNIATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
NEOPLASM RECURRENCE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 5 (6)
EPILEPSY (Nervous system disorders) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temozolomide Radiation (N=42) | Temozolomide Alone, Then Temozolomide Radiation (N=52)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 3 (5)
NAUSEA (Gastrointestinal disorders) | 13 (26) | 7 (8)
VOMITING (Gastrointestinal disorders) | 12 (15) | 4 (4)
GAIT DISTURBANCE (General disorders) | 3 (3) | 0 (0)
PYREXIA (General disorders) | 5 (5) | 3 (3)
DECREASED APPETITE (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
DIZZINESS (Nervous system disorders) | 0 (0) | 4 (4)
EPILEPSY (Nervous system disorders) | 1 (1) | 4 (5)
HEADACHE (Nervous system disorders) | 10 (12) | 2 (2)
INTRACRANIAL PRESSURE INCREASED (Nervous system disorders) | 0 (0) | 3 (7)
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institution and Principal Investigator (PI) have the right to publish/present study results. PI and Institution agree not to publish/present any interim study results. PI and Institution further agree to provide 30 days written notice to Sponsor prior to submission for publication or presentation to permit Sponsor to review drafts of abstracts and manuscripts for publication which report any study results. Sponsor shall have the right to review and comment on any Public Presentation.